CLINICAL TRIAL: NCT05739019
Title: A Prospective Observational Study of the Impact of a Recent Past COVID-19 Infection on the Live Birth Rates of Frozen Embryo Transfer Cycles
Brief Title: The Impact of Past Coronavirus Disease 19 (COVID-19) Infection on the Live Birth Rates of Frozen Embryo Transfer Cycles
Status: Completed | Type: Observational
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Other Study IDs: JIAI 2023-01
Record Dates: First submitted 2023-02-21; First posted 2023-02-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Frozen Embryo Transfer
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample is obtained on the day of progesterone supplementation day or luteinizing hormone surge day, and saved for further COVID-19 antibody test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19 infection group: Infertile women attending for frozen embryo transfer with a recent past COVID-19 infection
  Interventions: Other: frozen embryo transfer
- Control group: Infertile women attending for frozen embryo transfer without a recent past COVID-19 infection
  Interventions: Other: frozen embryo transfer

INTERVENTIONS:
Other: frozen embryo transfer — transfer one or two embryos in frozen embryo transfer cycles

SUMMARY:
This is a prospective observational study. In this study, we aim to investigate the effect of a recent past Covid-19 infection on the live birth rate in the frozen embryo transfer cycles

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-42 years at the time of ovarian stimulation for in vitro fertilization
2. Women have embryos frozen prior to COVID infection.

Exclusion Criteria:

1. Previous COVID infection before oocyte retrieval
2. Recipient of oocyte donation
3. Undergoing preimplantation genetic testing
4. Presence of hydrosalpinx or endometrial polyp which is not surgically treated

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women for frozen embryo transfer will be recruited for study after explanation and counseling if they fulfil the inclusion criteria and do not have the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
live birth rate | a live birth after 22 weeks gestation
  live birth rate of the frozen embryo transfer cycle (>22 weeks of gestation)

SECONDARY OUTCOMES:
serum hCG level | a blood pregnancy test is performed 14 days after the embryo transfer
  serum hCG level
clinical pregnancy | presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy
  presence of intrauterine gestational sac on ultrasound
ongoing pregnancy | viable pregnancy beyond gestation 12 weeks
  viable pregnancy beyond gestation 12 weeks
biochemical pregnancy | positive blood pregnancy test not followed by clinical pregnancy during 12 weeks gestation
  positive blood pregnancy test not followed by clinical pregnancy
implantation rate | number of gestational sacs per embryo transferred during 4 weeks of pregnancy
  number of gestational sacs per embryo transferred
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks
  more than one intrauterine sacs on scanning
ectopic pregnancy | ectopic pregnancy during 12 weeks gestation
  pregnancy outside the uterine cavity
miscarriage | the loss of a pregnancy before 22 weeks gestation
  the loss of a pregnancy before 22 weeks gestation
birth weight | a live birth after 22 weeks gestation
  birth weight of the baby delivered
serum COVID-19 antibody level | 7 days before embryo transfer
  serum COVID-19 antibody level immunoglobulin G and immunoglobulin M

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, PhD, Study Director — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared. Data will be available when beginning 3 months and ending 5 years following article publication. To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with.Data will be made available by the following way. Proposals should be directed to lihe198900@163.com. And data are available for 5 years at a third party website (link to be included after the article publication
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Lukassen S, Chua RL, Trefzer T, Kahn NC, Schneider MA, Muley T, Winter H, Meister M, Veith C, Boots AW, Hennig BP, Kreuter M, Conrad C, Eils R. SARS-CoV-2 receptor ACE2 and TMPRSS2 are primarily expressed in bronchial transient secretory cells. EMBO J. 2020 May 18;39(10):e105114. doi: 10.15252/embj.20105114. Epub 2020 Apr 14. PMID 32246845
- [Background] Zou X, Chen K, Zou J, Han P, Hao J, Han Z. Single-cell RNA-seq data analysis on the receptor ACE2 expression reveals the potential risk of different human organs vulnerable to 2019-nCoV infection. Front Med. 2020 Apr;14(2):185-192. doi: 10.1007/s11684-020-0754-0. Epub 2020 Mar 12. PMID 32170560
- [Background] Vaz-Silva J, Carneiro MM, Ferreira MC, Pinheiro SV, Silva DA, Silva-Filho AL, Witz CA, Reis AM, Santos RA, Reis FM. The vasoactive peptide angiotensin-(1-7), its receptor Mas and the angiotensin-converting enzyme type 2 are expressed in the human endometrium. Reprod Sci. 2009 Mar;16(3):247-56. doi: 10.1177/1933719108327593. Epub 2009 Jan 22. PMID 19164480
- [Background] Henarejos-Castillo I, Sebastian-Leon P, Devesa-Peiro A, Pellicer A, Diaz-Gimeno P. SARS-CoV-2 infection risk assessment in the endometrium: viral infection-related gene expression across the menstrual cycle. Fertil Steril. 2020 Aug;114(2):223-232. doi: 10.1016/j.fertnstert.2020.06.026. Epub 2020 Jun 17. PMID 32641214
- [Background] Aizer A, Noach-Hirsh M, Dratviman-Storobinsky O, Nahum R, Machtinger R, Yung Y, Haas J, Orvieto R. The effect of coronavirus disease 2019 immunity on frozen-thawed embryo transfer cycles outcome. Fertil Steril. 2022 May;117(5):974-979. doi: 10.1016/j.fertnstert.2022.01.009. Epub 2022 Jan 10. PMID 35216833
- [Background] Youngster M, Avraham S, Yaakov O, Landau Rabbi M, Gat I, Yerushalmi G, Baum M, Maman E, Hourvitz A, Kedem A. The impact of past COVID-19 infection on pregnancy rates in frozen embryo transfer cycles. J Assist Reprod Genet. 2022 Jul;39(7):1565-1570. doi: 10.1007/s10815-022-02517-w. Epub 2022 May 7. PMID 35525900